CLINICAL TRIAL: NCT00828698
Title: Finnish-German Prospective, Observational Follow-up Study on Risk Assessment of Mortality After Myocardial Infarction
Brief Title: FINGER; Finland-Germany Myocardial Infarction Study
Acronym: FINGER
Status: Completed | Type: Observational
Sponsor: University of Oulu (Other)
Collaborators: Medical Council of the Finnish Academy of Science (Unknown); Finnish Foundation for Cardiovascular Research (Other); Bundesministerium für Bildung, Wissenschaft, Forschung und Technologie (Unknown); Kommission für Klinische Forschung (Unknown); German Research Foundation (Other)
Responsible Party: Professor Heikki V Huikuri, University of Oulu
Other Study IDs: Finger-96
Record Dates: First submitted 2009-01-23; First posted 2009-01-26 (Estimated); Last update posted 2009-01-26 (Estimated); Status verified 2009-01

CONDITIONS: Acute Myocardial Infarction
Keywords: Death, sudden; All cause mortality
MeSH Terms: conditions — Death, Sudden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA samples from Finnish subjects in the study have been retained.

GROUPS / COHORTS (1):
- Acute Myocardial Infarction patients
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
The purpose of this observational study is to find characteristics and risk stratification methods for identification of subjects who have increased risk of death, especially sudden cardiac death, after acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myocardial infarction
* Consent to the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients who have been hospitalized for acute myocardial infarction from Munich, Germany and Oulu, Finland
Sampling Method: Non-Probability Sample
Dates: Start 1996-01; Primary Completion 2000-01 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 10years

SECONDARY OUTCOMES:
Sudden cardiac death | 10 years

CONTACTS AND LOCATIONS:
Locations (2):
- Oulu University Hospital, Oulu, Finland
- Deutsches Herzzentrum, Munich, Germany

REFERENCES:
- [Result] Makikallio TH, Barthel P, Schneider R, Bauer A, Tapanainen JM, Tulppo MP, Perkiomaki JS, Schmidt G, Huikuri HV. Frequency of sudden cardiac death among acute myocardial infarction survivors with optimized medical and revascularization therapy. Am J Cardiol. 2006 Feb 15;97(4):480-4. doi: 10.1016/j.amjcard.2005.09.077. Epub 2005 Dec 22. PMID 16461041
- [Result] Bauer A, Kantelhardt JW, Barthel P, Schneider R, Makikallio T, Ulm K, Hnatkova K, Schomig A, Huikuri H, Bunde A, Malik M, Schmidt G. Deceleration capacity of heart rate as a predictor of mortality after myocardial infarction: cohort study. Lancet. 2006 May 20;367(9523):1674-81. doi: 10.1016/S0140-6736(06)68735-7. PMID 16714188
- [Result] Makikallio TH, Barthel P, Schneider R, Bauer A, Tapanainen JM, Tulppo MP, Schmidt G, Huikuri HV. Prediction of sudden cardiac death after acute myocardial infarction: role of Holter monitoring in the modern treatment era. Eur Heart J. 2005 Apr;26(8):762-9. doi: 10.1093/eurheartj/ehi188. Epub 2005 Mar 18. PMID 15778204
- [Result] Peltola M, Tulppo MP, Kiviniemi A, Hautala AJ, Seppanen T, Barthel P, Bauer A, Schmidt G, Huikuri HV, Makikallio TH. Respiratory sinus arrhythmia as a predictor of sudden cardiac death after myocardial infarction. Ann Med. 2008;40(5):376-82. doi: 10.1080/07853890701884659. PMID 18499938